CLINICAL TRIAL: NCT06117592
Title: Co-design of Acute Oncology Standardised Assessment Documents and Their Evaluation
Brief Title: The CASCADE Project
Acronym: CASCADE
Status: Not yet recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: cftsp227
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Intervention: Retrospective data collection for pre-education intervention period: 1st April 2023- 1st June 2023
  Interventions: Other: Education, training and assessment intervention
- Post-Intervention: Retrospective data collection for post-education intervention period: 1st October 2023- 31st December 2023
  Interventions: Other: Education, training and assessment intervention

INTERVENTIONS:
Other: Education, training and assessment intervention — Staff competence assessment documents for acute oncology knowledge and skills

SUMMARY:
People with cancer, treated for cancer, or have been recently treated for cancer are at a higher risk of becoming rapidly unwell. This is referred to as an oncological emergency and can be life-threatening.

The investigators want to see if a new, standardised assessment of acute oncology knowledge and skills of all health care staff (The Acute Oncology Passport) following education and training, has an effect on the diagnosis and treatment of two relatively-common oncological emergencies: sepsis and MSCC? Sepsis is blood poisoning, which causes serious injuries if it is not diagnosed and treated as an emergency and may result in death if not treated quickly enough. MSCC is metastatic spinal cord compression, where the cancer presses on the spinal cord and can cause permanent paralysis. The investigators have chosen these two conditions, not only because of how serious and relatively common they are for people living with cancer, but also because all NHS Trusts in the UK routinely collect and report standardised data about patients who are admitted with suspected sepsis or MSCC.

The investigators plan to compare data that is routinely collected about the diagnosis and treatment of patients with suspected sepsis and MSCC before and after education, training and assessment of staff about acute oncology. The investigators will conduct 'secondary analysis' on the data, as it was originally collected for another purpose. The routinely data collected at five hospital Trusts across the UK from 1st April 2023 to 30th June 2023 and 1st October to 31st December 2023 will be included in this study.

This research is part of a larger UK-wide project, funded until March 2024 by NHS England Workforce, Training and Education Directorate. If acute oncology education, training and assessment of staff is shown to make a difference to patient diagnosis and treatment, the Acute Oncology Passports will be rolled-out nationally.

ELIGIBILITY:
Inclusion Criteria:

* All patient KPI's of interest that occur in the study time frame will be collected.

Exclusion Criteria:

* KPI data collected from people under the age of 18 KPI data other than items stated in this application, i.e. data that is not reporting neutropenic sepsis nor MSCC outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with suspected neutropenic sepsis or MSCC
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
Acute Oncology Key Performance Indicators (KPIs) | 1st April 2023- 31st December 2023
  These are routinely collected metrics by acute oncology teams for patients presenting with suspected neutropenic sepsis or metastatic spinal cord compression.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Griffin, PhD, Study Director — The Christie NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No